CLINICAL TRIAL: NCT05546437
Title: A Multicenter Retrospective Review to Evaluate the Feasibility of Dye Marking Using the Ion Endoluminal System
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-ION-R02
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects with Ion Endoluminal dye marking of pulmonary nodule for resection: Subjects in which a pulmonary lesion dye marking procedure was attempted or performed with the Ion Endoluminal System in anticipation of resection of the lesion
  Interventions: Device: Ion Endoluminal System

INTERVENTIONS:
Device: Ion Endoluminal System — Ion Endoluminal dye marking procedure for pulmonary nodule

SUMMARY:
The overall objective of this study is to assess the ability of the Ion Endoluminal System to perform pleural based tissue dye marking in anticipation of a lung resection.

DETAILED DESCRIPTION:
This study is a retrospective multicenter chart review of patients who underwent a pleural based tissue dye marking with the Ion Endoluminal System in anticipation of lung resection. The aim of the study is to assess the feasibility of the Ion Endoluminal System to perform pleural based tissue marking. As this is a retrospective study, the Ion dye marking procedure will have been performed according to the physician's standard technique. All consecutive cases in which a dye marking procedure was attempted and/or completed with the Ion Endoluminal System will be included.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older at the time of the procedure.
* Dye marking attempted/performed using the Ion Endoluminal Platform

Exclusion Criteria:

* Resection not performed following dye marking procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent an Ion Endoluminal dye marking procedure with a pulmonary nodule, 18 years or older, who subsequently underwent a resection of their pulmonary nodule.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Successful dye injection | Intra-procedure through the release of the final pathology report, approximately 3 days post-procedure
  The ability of the investigator to localize the marked lesion during resection, assessed by successful injection of dye, localization of due within the targeted area, and the ability to visualize the dye marking intra-operatively or on resected sample
Pneumothorax | Intra-procedure
  Incidence of all pneumothoraces related to the Ion procedure

SECONDARY OUTCOMES:
Adverse events | Intra-procedure until the start of the resection procedure
  All adverse events related to the Ion procedure
Procedure time | Intra-procedure
  Time from start of Ion dye marking procedure (defined as when the Ion catheter crosses the endotracheal tube [ETT]) to end of Ion dye marking procedure (defined as when the Ion catheter leaves the ETT).
Operative time | Intra-operative
  Time from start of resection procedure to end of resection procedure (skin-to-skin time)
Type of resection planned and performed | Intra-operative
  The type of resection procedure planned (ex., lobectomy, wedge resection) and whether that plan was altered after the dye marking procedure or resection has started.
Conversion to alternate approach or termination of procedure due to localization issues | Intra-operative
  Rate of resections converted to an alternative approach or terminated. Conversion is defined as a change in the procedural approach (either a different technology [ex., open resection] after the resection procedure has started. Termination is defined as prematurely ending the operation before the resection has been performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No